CLINICAL TRIAL: NCT03889288
Title: Innovative Device for Pain Management by Millimeter Band Radiation: Electronic-Pain Killer: First in Human Evaluation in Perioperative With Regard to a Control Group
Brief Title: Innovative Device for Pain Management by Millimeter Band Radiation: Electronic-Pain Killer
Acronym: EPIKARD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Remedee SA (Industry); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC18.170
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Aortic Valve Replacement
Keywords: pain treatment; intensive care; cardiology; medical device
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional management of postoperative pain (No Intervention): Patients who have had an aortic valve replacement surgery have a conventional management of pain after surgery. The pain is treated by morphine using a patient-controlled analgesia for the administration. Patients are recruiting prospectively or possibly retrospectively. The management is usual, nothing from the conventional care of patients change, only data will be collected.
- Medical device - electronic-pain killer (Experimental): In addition to the conventional management of postoperative pain, patients benefit from perioperative treatment sessions with medical device. Patients are recruiting prospectively.
  Interventions: Device: Medical device - electronic-pain killer

INTERVENTIONS:
Device: Medical device - electronic-pain killer — Treatment sessions with the medical device (no-marked EC): 2 sessions before surgery and 4 or 5 sessions until 48 hours after surgery. Each treatment sessions takes 45 minutes. Each session is spaced by 12 +/-3 hours.
  Arms: Medical device - electronic-pain killer

SUMMARY:
The objective of this study is to evaluate a new medical device in the management of pain. The principle of this new treatment is based on the emission of electromagnetic radiation in millimeter band. This new modality of pain management is evaluated in a perioperative management in patients undergoing surgery for aortic valve replacement.

The hypothesis is that the use of this medical device in perioperative would reduce the consumption of postoperative morphine with an identical quality of analgesia. The decline in morphine consumption would allow a decrease in opioid adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* candidate for an aortic valve replacement with extra-corporal flow.
* wrist size between 14.5 and 18.5 centimeters (for the experimental group)
* patient affiliated to social security
* signature of the informed consent (for the experimental group)

Exclusion Criteria for the control group :

* patient with diabetes
* patient with an evolutive cancer
* patient with cardiac assistance
* patient under the influence of opioid in the 48 hours before the surgery
* patient deprived of liberty by judicial or administrative decision
* patient subject to legal protection or unable to express his consent (guardianship or curators)

Exclusion Criteria for the experimental group :

* patient with diabetes
* patient with an evolutive cancer
* patient with surgery planning within 48 hours
* patient with cardiac assistance
* patient under the influence of opioid in the 48 hours before the surgery
* patient suffering from a dermatological disease such as oozing dermatitis, hyper sweating, or an unhealed lesion in the wrists.
* patient who has a piercing in the wrist or another metal material
* patient known for having a multi-resistant bacterial strain
* protected person referred to in Articles L1121-5 to L1121-8 of the Code of Public Health
* exclusion period of another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative consumption of morphine auto-administered in the experimental group in the first 48 hours : descriptive analysis | 48 hours
  The morphine cumulative consumption administered by auto-analgesia in the experimental group at 24 and 48 hours after the surgery

SECONDARY OUTCOMES:
Cumulative consumption of morphine auto-administered in the control group in the first 48 hours : descriptive analysis | 48 hours
  The morphine cumulative consumption administered by auto-analgesia in the control group at 24 and 48 hours after the surgery
Determine the number of patients required to demonstrate a 30% decrease in morphine consumption within the first 48h following aortic valve replacement surgery in a population treated with "Electronic-Pain-Killer" compared to conventional pain management | 48 hours
  Cumulative morphine consumption in milligrams, administered by auto-analgesia, at 48 hours post-operatively in the experimental and control groups.
Troponin's peak characterization in the first 48 hours postoperatively. | 48 hours
  The troponin is assessed in ng/ml in the two groups from the end of the surgery until 48 hours postoperatively
The Pain characterization: Echelle Numérique Standard; standard digital scale | 48 hours
  The patient pain is evaluated using the ENS (Echelle Numérique Standard; standard digital scale, score between 0 to 10) for both groups.
The hospitalization length in the intensive care unit | 48 hours
  For the two groups, the hospitalization length in the intensive care unit is assessed in hours.
Characterization of analgesic drugs | 48 hours
  The analgesic drugs are characterized by their class, dose and number of dose taken in the two groups since they are in the intensive care unit.
Number of postoperative nausea or vomiting events (number of PONV) in the experimental group | 48 hours
  In the experimental group, the number of PONV events requiring a treatment is assessed.
Delirium events in the experimental group | 48 hours
  The number of delirium events is assessed using the CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) scale in the experimental group.
Adverse effect from the medical device | 48 hours
  The number of adverse effects from the medical device is assessed from the first session with the medical device to the follow-up visit.
Description of the medical device use | 48 hours
  Log files of the medical device are extracted. The length of each session, the start and end session times, each stopping is analysed.
Medical device acceptability : score | 48 hours
  This score has been specifically created for the electronic pain killer medical device. Each item range from 0 (the worst) to 10 (the best).
Medical device acceptability : descriptive analysis | 48 hours
  Open questions will be asked in a questionnaire without scale. A descriptive analysis will be done with the answers.
Use Error evaluation : System Usability Scale (SUS) | 48 hours
  The System Usability Scale (SUS) contains 10 questions that are rated on a scale from 1 to 5. "The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100." Jeff Sauro established the average score of SUS is 68.
  The score can go from 0 (worst) to 100 (best).
Subgroup analysis excluding patients who have had Nefopam administration | 48 hours
  To avoid a potential bias confusion, patients taking Nefopam drug are excluded from the analyses and all the previous outcome are assessed again.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Albaladejo, MD, PhD, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, France